CLINICAL TRIAL: NCT06318923
Title: Social and Moral Cognition in Multiple Sclerosis
Acronym: COSMOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC-P00117
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Neuropsychological Tests; Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple sclerosis patients (Other): MS patients with the relapsing-remitting form (RRMS) and Expanded Disability Status Scale (EDSS) ≤ 4
  Interventions: Other: Socio-demographic questionnaire, moral judgment task, cognitive tests, psychoaffective assessment; Other: MS questionnaire
- Control participants (Other): Patients without global cognitive impairment
  Interventions: Other: Socio-demographic questionnaire, moral judgment task, cognitive tests, psychoaffective assessment; Other: MONTREAL COGNITIVE ASSESSMENT (MoCA) test

INTERVENTIONS:
Other: Socio-demographic questionnaire, moral judgment task, cognitive tests, psychoaffective assessment — The demographic questionnaire collects demographic information: gender, age, level of education, laterality, history of psychiatric or neurological disorders.
  The moral judgment task consists in completing 20 vignettes of moral dilemmas. Cognitive disorders will be assessed using the Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) battery. If the patient has taken the BICAMS battery recently (less than 6 months), and with no change in pathology since then, the results of these tests will be used in this study.
  Affective disorders will be assessed using the following tests:
  * The Beck Depression Inventory-Fast Screen (BDI-FS) to assess the level of depression,
  * State trait anxiety inventory-Y (STAI-Y) to assess anxiety,
  * Toronto Alexithymia Scale-20 (TAS-20)to assess alexithymia,
  * The Empathy Quotient-8 (EQ-8) to assess participants' level of empathy,
  * The Dot Probe Task to assess participants' emotional information processing style.
Other: MS questionnaire — This questionnaire collects key information on the participant's pathology: clinical form, date of first symptoms, diagnosis, last attack, as well as latest EDSS and functional scores.
  Arms: Multiple sclerosis patients
Other: MONTREAL COGNITIVE ASSESSMENT (MoCA) test — The MoCA is a screening tool for neurocognitive impairment, designed primarily to detect milder impairment. The MoCA is a short-answer questionnaire that includes a number of tasks to be completed by the individual. The items assessed are grouped into six subsections: short-term memory, visuospatial skills, executive functions, attention, concentration, working memory, language and orientation in time and space. The tests proposed are often more complex than those found in the mini-mental state examination (MMSE).
  Arms: Control participants

SUMMARY:
Multiple Sclerosis (MS) is a chronic, progressive disease that affects young adults (aged between 20 and 40) and has a major impact on patients' quality of life. Cognitive disorders in MS are common, affecting 40-60% of patients. Among these disorders, the presence of social cognition disorders is common. Within social cognition, the moral judgment has been an object of research in order to understand the determinants of moral decision-making: how and why individuals make moral choices with regard to a set of prescriptions and social norms. Compared to control subjects, MS patients show a decrease in moral permissiveness, as well as an increase in moral relativity and emotional reactivity. Thus, it would seem that MS patients issue more deontological choices (lower moral permissiveness). Given that these patients also exhibit empathy deficits and higher alexithymia, these patterns are surprising. Indeed, in other clinical populations, low empathic abilities and high alexithymia are linked to utilitarian rather than deontological moral judgments.

The objective of this project is to analyze the process of decision-making carried out by patients during moral dilemma situations in comparison with control individuals and verify whether the presence of a positivity bias could explain the more deontological choices made by some patients. Indeed, some work has shown that older individuals make more deontological moral judgments than younger adults. These results are also observed with young individuals when their future temporal perspectives have been experimentally constrained.

DETAILED DESCRIPTION:
Among the explanatory factors of interest, motivational factors (future temporal perspectives and emergence of a positivity bias), as well as cognitive and affective factors (by means of neuropsychological assessment) and neurophysiological factors (by means of electrodermal response) will be investigated.

From a clinical point of view, a change in decision-making concerning choices with a strong emotional valence can have an impact on patients' daily lives and their course of care. Indeed, MS patients regularly have to make crucial choices about their treatment and care. A modification of decision-making patterns in these situations would represent a major challenge. A good understanding of these patterns will thus contribute to the development of appropriate management procedures to mitigate the impact on patients' daily lives.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 to 55.
* Understanding and able to express themselves in French.
* Characteristics according to groups:
* MS patient group:

  * relapsing-remitting form (RRMS)
  * with EDSS ≤ 4
  * with no significant motor, cerebellar or somesthesic disorders of the upper limbs or visual disorders (specific EDSS parameter ≤ 2)
  * absence of relapse in the last 6 weeks
* Control groups:

  * absence of known global cognitive deterioration.
* Understanding and signing of the informed consent and information letter concerning participation in the study.
* Beneficiary of health insurance coverage.

Exclusion Criteria:

* People with previous neurological pathologies, head trauma with loss of consciousness, known psychiatric pathologies (excluding anxiety-depressive syndrome), serious general illnesses, perceptual or dysarthric disorders preventing verbal communication or reading,
* Severe cognitive impairment in MS patients, i.e. an SDMT score < -2.5 if the BICAMS battery is present in the patient's file and is less than 6 months old.
* Severe depressive syndrome, with a BDI-FS score > 10
* People with sensory disorders (visual and auditory) that interfere with neuropsychological testing;
* Major sensory disorders or cerebellar syndrome
* Sensory deficits (visual or auditory)
* Treatment with psychotropic drugs
* Adults under guardianship, curatorship, persons deprived of liberty.
* Pregnant or breast-feeding women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Moral dilemma judgments | 3 hours
  The measure will be carried out using a series of 20 vignettes.These vignettes present different scenarios of fictional moral dilemmas, and the subject must make a choice. This test therefore results in 20 binary measures, which can be separated according to the type of scenario.
  In this task, for each vignette, the type of choice made is measured, along with levels of moral permissibility, subjective emotional reactivity and moral relativity.
  For this scale:
  Type of choice: binary yes/no (utilitarian/deontological) ; reflects an answer type (no better or worse outcome) Moral permissibility: Likert Scale from 0 to 10 ; reflects an answer type (no better or worse outcome) Subjective emotional reactivity : Likert Scale from 0 to 10 ; reflects an answer type (no better or worse outcome) Subjective emotional r

SECONDARY OUTCOMES:
Explicit time perspective inventory test | 3 hours
  Participants indicate, on scales ranging from 1 (not at all) to 5 (completely) their levels of agreement on 10 items assessing their future time perspective (e.g. "I plan to set many new goals for myself in the future"). A total score is extracted.
Implicit time perspective inventory test | 3 hours
  Participants are presented with 20 fill-in-the-blank words. These words can be completed either with words referring to future time ("target words"), or with neutral words. The percentage of target words is extracted.
Dot Probe Task | 3 hours
  This task allows us to assess whether individuals tend to pay more attention to positive or negative information. During the dot-probe task, participants are situated in front of a computer screen and asked to stare at a fixation cross on the center of the screen. Two stimuli, one of which is neutral and one of which is threatening, appear randomly on either side of the screen. The stimuli are presented for a predetermined length of time (most commonly 500ms), before a dot is presented in the location of one former stimulus. Participants are instructed to indicate the location of this dot as quickly as possible, either via keyboard or response box. Latency is measured automatically by the computer. The fixation cross appears again for several seconds and then the cycle is repeated. Quicker reaction time to the dot when it occurs in the previous location of a threatening stimulus is interpreted as vigilance to threat.
Level of moral permissibility | 3 hours
  This test aims to measure to what extent the participant finds the proposed solution acceptable. For example: How acceptable do you find it to activate the switch in this situation? An 11-point Likert scale is displayed, ranging from "Not at all" to "Absolutely".
Level of emotional reactivity | 3 hours
  This test aims to measure the individual's emotional (subjective) reaction to a moral dilemma. For example: What emotion does this situation arouse in you? An 11-point Likert scale is displayed, ranging from "None" to "Intense emotion".
Moral relativity level | 3 hours
  This test aims to measure to what extent the participant feels this choice is consensual. For example: Out of 100 people who responded to this scenario, how many would answer as you do? An 11-point Likert scale is displayed below the question, ranging from 0% to 100%.
Brief International Cognitive Assessment for Multiple Sclerosis | 3 hours
  This test enables the assessment of cognitive disorders. The battery's 3 component tests are as follows:
  * California Verbal Learning Test (CVLT): This test is based on a master list of 16 words belonging to 4 distinct semantic categories . The list is presented 5 times, with the patient asked to recall it immediately after each presentation and after a 20-minute delay. A main score is extracted.
  * Brief Visuo-spatial Memory Test (BVMT): This test involves 6 simple geometric drawings. 3 presentation/recall phases follow one another, during which the patient is shown the sheet for 10 seconds, followed by an immediate recall phase. A delayed recall phase (at 7 minutes) is also proposed. A main score is extracted.
  * Symbol Digit Modalities Test (SDMT): a coding test in which the patient has 90 seconds to orally state the correspondence of digits (from 1 to 9) to 9 different symbols (matched according to a correspondence standard). The number of correct answers is measured.
The Beck Depression Inventory | 3 hours
  This is a 21-question multiple-choice self-report inventory, for measuring the severity of depression.
  When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity. The standard cut-off scores are as follows:
  0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression. Higher total scores indicate more severe depressive symptoms.
State-Trait Anxiety Inventory | 3 hours
  The State-Trait Anxiety Inventory is one of the first tests to assess both state and trait anxiety separately. Each type of anxiety has its own scale of 20 different questions that are scored.[10] Scores range from 20 to 80, with higher scores correlating with greater anxiety.
Toronto Alexithymia Scale (TAS)-20 | 3 hours
  The TAS-20 is a self-report scale that is comprised of 20 items. Items are rated using a 5-point Likert scale whereby 1 = strongly disagree and 5 = strongly agree. There are 5 items that are negatively keyed (items 4, 5, 10, 18 and 19). The total alexithymia score is the sum of responses to all 20 items, while the score for each subscale factor is the sum of the responses to that subscale. The TAS-20 uses cutoff scoring: equal to or less than 51 = non-alexithymia, equal to or greater than 61 = alexithymia. Scores of 52 to 60 = possible alexithymia.
Empathy quotient-8 (EQ-8) | 3 hours
  This is an 8-item self-questionnaire. Subjects are asked to self-assess their level of empathy by positioning themselves, for each item, on a rating scale from 1 to 5 (1 = completely disagree and 5 = completely agree). The total score is analyzed.
Electrodermal response | 3 hours
  During performance of the moral judgment task, an electrodermal response recording device will be installed via two electrodes placed on the participant's non-dominant hand to measure objective emotional reactivity. Individuals' signals are examined in relation to their own baseline levels (without stimuli, Baseline measure), which will serve as a reference for interpreting the signals obtained during the task.

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice DEGRAEVE, Principal Investigator — Catholic University of Lille Faculty of Letters and Humanities
Locations (2):
- France (2):
  - Hôpital Saint-Vincent-de-Paul - Neurologie, Lille
  - Hôpital Saint-Philibert - Neurologie, Lomme

IPD SHARING:
Plan to Share IPD: No